CLINICAL TRIAL: NCT04058301
Title: Text-Enabled Ascertainment and Community Linkage for Health
Acronym: TEACH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Margaret Samuels-Kalow, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019P001579
Record Dates: First submitted 2019-05-17; First posted 2019-08-15 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Emergency Medicine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handout (No Intervention): Participants receive a generic handout about resources in Boston
- Text message (Experimental): Participants receive a generic handout about resources in Boston and a text message with a geographically proximate resource
  Interventions: Other: Text message information

INTERVENTIONS:
Other: Text message information — Geographically proximate resources delivered by text message
  Arms: Text message

SUMMARY:
The goal of this study is to pilot test a novel tool for health related social needs screening and linkage to community resources in the ED by randomizing participants to standard handout v. handout + text message with resource information.

ELIGIBILITY:
Inclusion Criteria:

* 51 ZIP codes included in our database of community resources ("catchment area")
* >=18 years old
* plan for discharge home
* speak either English or Spanish
* live within the catchment area for the study
* have a cellphone with text messaging capabilities
* ability to respond to text messages from the study team.

Exclusion Criteria:

* Patients who are intoxicated
* on a Section 12
* lack capacity to consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction: Likert scale | 3-5 days
  Participants will be asked about their satisfaction with the program measured on a Likart scale. Options will include "Extremely or Quite a bit; Somewhat; A little bit or Not at all"

SECONDARY OUTCOMES:
Resource use | 3-5 days
  Participants will be asked about actual and planned resource use
Health status | 3-5 days
  Participants will be asked about health status. In general, how would you rate your health? Excellent, Very good, Good or Fair,Poor

OTHER OUTCOMES:
ED utilization | 30 days
  Chart review of ED visits and potentially preventable utilization

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No